CLINICAL TRIAL: NCT03546361
Title: A Phase I Trial of Intratumoral Administration of CCL21-Gene Modified Dendritic Cell (Ad-CCL21-DC) Combined With Intravenous Pembrolizumab for Advanced NSCLC
Brief Title: CCL21-Gene Modified Dendritic Cell Vaccine and Pembrolizumab in Treating Patients With Stage IV Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other); Merck Sharp & Dohme LLC (Industry); LUNGevity Foundation (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17-000174; NCI-2018-01244 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HEMONC CIRM IST Lung (Other: UCLA / Jonsson Comprehensive Cancer Center); K08CA245249 (NIH)
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Ad-CCL21-DC vaccine, pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes followed by autologous dendritic cell-adenovirus CCL21 vaccine by CT-guided or bronchoscopic IT injection on days 0, 21, and 42. Patients then receive pembrolizumab every 3 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Autologous Dendritic Cell-Adenovirus CCL21 Vaccine; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Autologous Dendritic Cell-Adenovirus CCL21 Vaccine — Given via CT-guided or bronchoscopic IT injection
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase I trial studies the side effects and best dose of autologous dendritic cell-adenovirus CCL21 vaccine (CCL21-gene modified dendritic cell vaccine) combined with intravenous pembrolizumab, and to see how well they work in treating patients with stage IV non-small cell lung cancer. Vaccines made from a gene-modified virus may help the body build an effective immune response to kill tumor cells. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of tumor cells to grow and spread. Giving CCL21-gene modified dendritic cell vaccine with pembrolizumab may work better in treating patients with stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Dose escalation: To determine the safety and maximum tolerated dose (MTD) of intratumoral injection of autologous dendritic cell-adenovirus CCL21 vaccine (CCL21 gene-modified DC [Ad-CCL21-DC]) when combined with intravenous pembrolizumab in 1) patients with advanced non-small cell lung cancer (NSCLC) without a sensitizing epidermal growth factor receptor (EGFR) mutation and/or anaplastic lymphoma kinase (ALK) gene rearrangement who have received prior systemic anti-cancer therapy for advanced disease that includes a PD -1 and/or PD-L1 inhibitor or 2) patients who have sensitizing EGFR mutations and/or ALK gene rearrangements and have received prior tyrosine kinase inhibitor therapy.

II. Dose expansion: To evaluate the objective response rate (ORR) in subjects treated with the dose established during dose escalation (ExD) of intratumoral injection of Ad-CCL21-DC when administered with intravenous pembrolizumab in 1) patients with advanced non-small cell lung cancer (NSCLC) without a sensitizing epidermal growth factor receptor (EGFR) mutation and/or anaplastic lymphoma kinase (ALK) gene rearrangement who have received prior systemic anti-cancer therapy for advanced disease that includes a PD -1 and/or PD-L1 inhibitor or 2) patients who have sensitizing EGFR mutations and/or ALK gene rearrangements and have received prior tyrosine kinase inhibitor therapy.

SECONDARY OBJECTIVES:

I. To define the adverse event (AE) profile of intratumoral injection of Ad-CCL21-DC (determined during dose escalation) when administered with intravenous pembrolizumab in 1) patients with advanced non-small cell lung cancer (NSCLC) without a sensitizing epidermal growth factor receptor (EGFR) mutation and/or anaplastic lymphoma kinase (ALK) gene rearrangement who have received prior systemic anti-cancer therapy for advanced disease that includes a PD -1 and/or PD-L1 inhibitor or 2) patients who have sensitizing EGFR mutations and/or ALK gene rearrangements and have received prior tyrosine kinase inhibitor therapy.

II. To determine drug target activity by analyzing serial pre- and post-treatment biopsies and blood specimens of intratumoral injection of Ad-CCL21-DC (determined during dose escalation) when administered with intravenous pembrolizumab in 1) patients with advanced non-small cell lung cancer (NSCLC) without a sensitizing epidermal growth factor receptor (EGFR) mutation and/or anaplastic lymphoma kinase (ALK) gene rearrangement who have received prior systemic anti-cancer therapy for advanced disease that includes a PD -1 and/or PD-L1 inhibitor or 2) patients who have sensitizing EGFR mutations and/or ALK gene rearrangements and have received prior tyrosine kinase inhibitor therapy.

OUTLINE: This is a dose-escalation study of autologous dendritic cell-adenovirus CCL21 vaccine.

Patients receive pembrolizumab intravenously (IV) over 30 minutes followed by autologous dendritic cell-adenovirus CCL21 vaccine by computed tomography (CT)-guided or bronchoscopic intratumoral (IT) injection on days 0, 21, and 42. Patients then receive pembrolizumab every 3 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at day 63 and every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically confirmed diagnosis of NSCLC will be enrolled in this study.
* Stage IV pathologically proven NSCLC.
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
* Must have received prior systemic anti-cancer therapy for advanced disease that includes either:

  * A PD-1 and/or PD-L1 inhibitor in patients without a sensitizing EGFR mutation and/or ALK gene rearrangement or.
  * Have received prior tyrosine kinase inhibitor therapy in patients with a sensitizing EGFR mutation and/or ALK gene rearrangement. For patients with sensitizing EGFR mutations, prior therapy must include osimertinib if a T790M mutation in the EGFR gene has been documented, and for patients with ALK gene rearrangements, prior therapy must include a second generation ALK inhibitor (e.g. alectinib, brigatinib, ceritinib). Note: For this group, prior cytotoxic chemotherapy is permitted, but prior therapy with a PD-1 or PD-L1 inhibitor is not permitted.
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1.
* Absolute neutrophil count (ANC) >= 1500/uL.
* Platelets >= 100,000/uL.
* Hemoglobin >= 9.0 g/dL or >= 5.6 mmol/L.

  * Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.
* Creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 30mL/min for participant with creatinine levels >1.5 x institutional ULN.

  * Creatinine clearance (CrCl) should be calculated per institutional standard.
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 x ULN.
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN (=< 5 x ULN for participants with liver metastases).
* International normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or activated partial prothrombin time (aPTT) is within therapeutic range of intended use of anticoagulants.
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants.
* A lesion that either:

  * Is intended to be accessed bronchoscopically OR.
  * Is intended to be accessed with computed tomography (CT) guided transthoracic injection and in the estimation of the radiologist performing the procedure will not require transversing a bullae that significantly increases the risk of pneumothorax.
* Male participants:

  * A male participant must agree to use a contraception of this protocol during the treatment period and for at least 4 months after the last dose of study treatment and refrain from donating sperm during this period.
* Female participants:

  * A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    * Not a woman of childbearing potential (WOCBP). OR
    * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 4 months after the last dose of study treatment.

Exclusion Criteria:

* Comorbid disease or a medical or psychiatric condition that would impair the ability of the patient to receive or comply with the study protocol.
* Any use of systemic corticosteroids within 10 days of treatment initiation.
* Respiratory failure (defined as oxygen saturation [SaO2] < 90% on room air; partial pressure of carbon dioxide [PCO2] > 45 mmHg; or forced expiratory volume in one second [FEV1] <1.0 liter).
* Acute viral, bacterial, or fungal infection, which requires specific therapy. Acute therapy must have been completed at least 7 days prior to study treatment.
* Human immunodeficiency virus (HIV) infected patients (defined as HIV-1/HIV-2 antibody positive).
* Patients with active hepatitis B or C. Active hepatitis B is defined as a known positive hepatitis B virus surface antigen (HBsAg) result. Active hepatitis C is defined by a known positive hepatitis (hep) C antibody (Ab) result and known quantitative hepatitis C virus (HCV) ribonucleic acid (RNA) results greater than the lower limits of detection of the assay.
* Hypersensitivity to any reagents used in the study.
* Pregnancy or inadequate contraception.
* Lactating females.
* Clinically active brain metastases, defined as untreated and symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms. In patients with brain metastases that have been treated with radiation therapy, treatment must end at least 14 days prior to starting study treatment. History of leptomeningeal disease is exclusionary regardless of prior therapy.
* Subjects with organ allografts.
* Previous or concurrent evidence of autoimmune disease requiring systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require inhaled steroid or local steroid injections will not be excluded from the study. Subjects with hypothyroidism who are managed by hormone replacement will not be excluded from the study.
* Patients with a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2026-01-11 (Estimated); Study Completion 2027-01-11 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD)/maximum administered dose (MAD) (dose escalation) | At 28 days
Overall response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 (dose expansion) | Up to 1 year
  Demographic characteristics of patients including age, gender ethnicity, performance status, prior therapies and other baseline characteristics as collected on the case report form will be summarized by Ad-CCL21-DC dose cohort using descriptive statistics. For continuous variables, descriptive statistics (n, mean, standard deviation, standard error, median, minimum, and maximum) will be provided. For categorical variables, patient counts and percentages will be provided. Categories for missing data will be presented if necessary. The ORR will be summarized using descriptive statistics by dose level. The ORR will be analyzed using one-sample exact Binomial test for the patients treated at MTD or MAD in both the dose escalation phase and dose expansion phase. The 95% exact confidence interval (CI) will be provided.

SECONDARY OUTCOMES:
Incidence of adverse events per Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 | Up to 1 year
Biomarker assessment | Up to 1 year
  Immunohistochemistry (IHC) will be conducted to assess biomarkers including PD-1, PD-L1, CD8, and CD4 (DC) expression. All immunologic parameters will be summarized using mean, standard deviation, median, percentile for continuous variables, and frequency and percentage for categorical variables. The summary statistics will be tabulated by time and dose level. Several plots, such as stem-and-leaf plot and normal probability plot, will be constructed to check the distribution of each variable. Transformation will be applied if the distribution of the variable is not normal. For the tumor tissue immune parameters measured at different time points, the post- treatment values will be compared with the pre-treatment values using either paired t-test or Wilcoxon signed-rank test. Box plots for pre-treatment and post-treatment data will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Edward B Garon, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States